CLINICAL TRIAL: NCT03271723
Title: The 2015 Pelotas (Brazil) Birth Cohort Study
Status: Completed | Type: Observational
Sponsor: Federal University of Pelotas (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Principal Investigator, MARLOS RODRIGUES DOMINGUES, PhD, Federal University of Pelotas
Other Study IDs: C2015
Record Dates: First submitted 2017-08-25; First posted 2017-09-05 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: Mother-Child Relations; Preterm Birth; Infant Development; Breast Feeding; Physical Activity; Pregnancy Related; Medicine, Narrative
Keywords: cohort studies; infant development; pregnancy; Brazil; observational studies; epidemiology; maternal health
MeSH Terms: conditions — Premature Birth; Breast Feeding; Motor Activity; Narrative Medicine | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational study — No intervention

SUMMARY:
This is the fourth birth cohort to be carried out in the city of Pelotas (Brazil) including more than 4 thousand children followed-up since the pre-natal period to study maternal-child health.

DETAILED DESCRIPTION:
The Pelotas 2015 Birth cohort is the fourth birth cohort being established in Pelotas since 1982. Data is being collected with a focus on maintaining fidelity to the tools and instruments used in the previous cohorts with minimal adaptations when necessary. All children born in Pelotas during 2015 were included in the cohort, and the cohort has been followed four times, at birth, 3, 12 and 24 months (ongoing). In addition, an antenatal study identified and interviewed 73.8% of the mothers that subsequently delivered children that are now part of the cohort. The 4275 children included in the cohort are part of extensive assessments that include information on antenatal health and care, pregnancy health, gestational age, physical activity, sleep, health behaviours, socio-demographic characteristics, perinatal conditions, child anthropometry, delivery information, child mortality and morbidity, nutrition, growth, breastfeeding, neuro-cognitive development, access to health services, medicine use by both mother and child and genetic material. The cohort also nests 2 randomized clinical trials and a series of sub-studies. The data is starting to be analyzed and, among other findings, confirm the already alarming trends in surgical deliveries, amounting to 65.2% of all deliveries in 2015.

ELIGIBILITY:
Inclusion Criteria:

* live births
* mothers living in urban area of the city
* delivered during 2015

Exclusion Criteria:

* stillbirths below 500g
* mothers living outside Pelotas

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All live births from mothers living in Pelotas during the year 2015 were included in the birth cohort to be followed-up since birth.
Sampling Method: Non-Probability Sample
Enrollment: 4275 (Actual)
Dates: Start 2014-04-15 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Preterm birth | At birth
  Births before 37 weeks of pregnancy

SECONDARY OUTCOMES:
Physical activity | Second trimester of pregnancy
  Physical activities performed during pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Pedro C Hallal, PhD, Principal Investigator — Federal University of Pelotas; Diego G Bassani, PhD, Principal Investigator — SickKids, Toronto; Mariângela F Silveira, PhD, Principal Investigator — Federal University of Pelotas; Andrea D Bertoldi, PhD, Principal Investigator — Federal University of Pelotas
Locations (1):
- Physical Education School, Pelotas, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Domingues MR, Bassani DG, da Silva SG, Coll Cde V, da Silva BG, Hallal PC. Physical activity during pregnancy and maternal-child health (PAMELA): study protocol for a randomized controlled trial. Trials. 2015 May 24;16:227. doi: 10.1186/s13063-015-0749-3. PMID 26003406
- [Background] Santos IS, Bassani DG, Matijasevich A, Halal CS, Del-Ponte B, da Cruz SH, Anselmi L, Albernaz E, Fernandes M, Tovo-Rodrigues L, Silveira MF, Hallal PC. Infant sleep hygiene counseling (sleep trial): protocol of a randomized controlled trial. BMC Psychiatry. 2016 Sep 2;16(1):307. doi: 10.1186/s12888-016-1016-1. PMID 27590170
- [Result] Coll CVN, da Silveira MF, Bassani DG, Netsi E, Wehrmeister FC, Barros FC, Stein A. Antenatal depressive symptoms among pregnant women: Evidence from a Southern Brazilian population-based cohort study. J Affect Disord. 2017 Feb;209:140-146. doi: 10.1016/j.jad.2016.11.031. Epub 2016 Nov 26. PMID 27914247
- [Result] Coll CV, Domingues MR, Hallal PC, da Silva IC, Bassani DG, Matijasevich A, Barros A, Santos IS, Bertoldi AD. Changes in leisure-time physical activity among Brazilian pregnant women: comparison between two birth cohort studies (2004 - 2015). BMC Public Health. 2017 Jan 25;17(1):119. doi: 10.1186/s12889-017-4036-y. PMID 28122524